CLINICAL TRIAL: NCT04494061
Title: A Clinical Study to Investigate Interferon Gamma (IFNɣ) Signature in Patients Post HSCT and in Patients With Impaired HSC Proliferation Pre-transplant
Status: Terminated | Type: Observational
Why Stopped: Decision related to Business Priorities, Assessment of Development Options
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: PRA Health Sciences (Industry); Cytel Inc. (Industry); BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: NI-0501-13
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Graft Failure
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HSCT - Hematopoetic Stem Cell Proliferation: Patients who received hematopoietic stem cell transplant
  Interventions: Procedure: blood collection
- IHSCP - Impaired HSC proliferation: Patients with impaired hematopoietic stem cell proliferation
  Interventions: Procedure: blood collection

INTERVENTIONS:
Procedure: blood collection — Blood samples will be collected as per protocol defined schedule. There is no investigation drug in this study.

SUMMARY:
Clinical study designed to collect blood for research purposes in patients after hematopoietic stem cell transplantation (HSCT) or in patients with a medical condition where the blood cells production is impaired. The blood samples will be used to study the role of Interferon gamma (IFNɣ) in graft failure or impairment of hematopoietic stem cell proliferation. The IFNɣ signature will be assessed by measuring primarily IFNɣ and C-X-C Motif Chemokine Ligand 9 (CXCL9).

DETAILED DESCRIPTION:
This clinical study is designed to investigate IFNγ activity in two cohorts of patients.

* First group will include patients post HSCT at risk of graft failure (GF) based on their underlying diseases and on the transplant procedure.
* Second group will contain patients with conditions where HSC proliferation is impaired (e.g. aplastic anemia) and with matched controls (healthy volunteers (HV) samples collected outside this clinical protocol).

IFNɣ activity will be assessed by measuring IFNγ and CXCL9 in serum.

For HSCT cohort, the following sampling time points are required: on day -7, pre HSCT on day 0, 1, 3, 5, 9, 13, 17, 21, 28, 31, 38 and one additional sample at the time when primary or secondary GF is suspected if not on the planned schedule. In addition, the following time points are recommended: day 7, 11, 15, 19, 24, 35, 42. It is also suggested to collect a sample when Graft vs Host Disease (GVHD) is diagnosed during any visit that the patients will attend as part of his/her standard treatment during the first 100 days post-transplant. The patient will be followed up until around day 100 post-transplant. This follow up will consist of capturing HSCT outcome information from patient hospital records around day 100.

For IHSCP cohort pre-transplant, it is recommended that, one sample per patient at the time of diagnosis (if possible not more than 1 week from the date of diagnosis) is collected. Age/sex matched control samples should be collected from healthy volunteers or patients with malignant disease outside of this protocol after appropriate consent.

Different sets of data will be collected for the HSCT and IHSCP cohorts respectively as described below:

Data collected for both cohorts

* Age and sex
* Inflammatory markers
* IFNɣ
* CXCL9
* Other potential relevant exploratory biomarkers
* Diagnosis
* Date of disease diagnosis
* Relevant medical history
* Date and time of sample collection

Data collected for HSCT cohort only

* Laboratory parameters assessed at the site laboratory on the date of sample collection and between collection dates when available:
* Absolute neutrophile count (ANC) and Platelets will be measured as per the schedule of assessment, if possible when routine monitoring of patient health is conducted
* Ferritin and Chimerism data will be collected when available (if measured as per site routine practice)
* Concomitant medications at the time of sample collection and between collection dates
* Presence of infection at the time of sample collection with the date of onset
* Presence of donor specific antibodies (DSA)
* Transplant information
* Date of start of conditioning
* Type of conditioning (Reduced Intensity Conditioning (RIC) / Myeloablative Conditioning (MAC) / Non-myeloablative Conditioning (NMAC) and medications
* Transplant details (donor type, degree of match, transplant manipulation, stem cell source)
* Date of transplant
* Date of primary / secondary GF or of confirmed engraftment
* GVHD with the date of onset
* Post-transplant treatment and date (Donor Lymphocyte Infusion (DLI), Stem Cell (SC) boost, growth factor, GVHD prophylaxis, second HSCT procedure)

Data collected for IHSCP cohort only

* Disease severity
* In addition, the following data will be recorded for pediatric patients up to 18 years old, if available:
* PNH clones
* History of hepatitis
* Karyotype

Study duration:

The study will be conducted, until the required number of patients is recruited.

* HSCT cohort: At patient level, the study will last about 100 days from pre-transplant blood collection to last follow up data collection around day 100 post HSCT, matching the standard HSCT patient care
* IHSCP cohort: At patient level the study will last 1 day.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to the use of their clinical data and biological samples for research investigations.
* In HSCT cohort:

  * Patients with underlying:

    i. non-malignant hematological disease (e.g. autoimmune and metabolic disorders, aplastic anemia, Sickle cell anemia, Fanconi anemia, Diamond-blackfan anemia, thalassemia, osteopetrosis, Wiskott-Aldrich syndrome, severe combined immunodeficiency) or ii. malignant disease with higher risk of GF, i.e. Acute Myeloid Leukemia (AML) and Acute Lymphoblastic Leukemia (ALL) with primary induction failure, second partial remission or relapse; Chronic Myeloid Leukemia (CML) in blastic phase (circulating blast or blast above 5% in biopsy); Non Hodgkin and Hodgkin Lymphoma and multiple myeloma with primary induction failure, second partial remission or relapse, myelodysplastic syndromes (MDS) and myeloproliferative disorders (MPD) with splenomegaly, myelofibrosis with portal hypertension pre-transplant, MDS/MPD overlap syndromes
  * and who received allogeneic HSCT and are at higher risk of graft failure based on at least one of the following criteria: i. Having received reduced intensity conditioning (RIC) or non myeloablative conditioning (NMA) combined with a non-malignant disease or having received graft from Bone Marrow (BM) ii. Ex vivo T cell depleted graft iii. Graft from mismatched unrelated donor or haploidentical donor iv. Graft from Umbilical Cord Blood (UCB)
* In the IHSCP cohort:

  * Patients with IHSCP pre-transplant (e.g. aplastic anemia)

Exclusion Criteria:

* HLH patients
* Body weight < 10kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients post HSCT at risk of graft failure based on their underlying diseases and on the transplant procedure.
  * Patients with conditions where HSC proliferation is impaired (e.g. aplastic anemia) and with respective controls (healthy volunteers (HV)).
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
HSCT cohort: IFNγ signature pre-and post-transplant | Day (-7) to day 100
  IFNγ, CXCL-9 and exploratory biomarkers in serum samples
HSCT cohort: Relationship between IFNγ and the risk of graft failure | Day (-7) to day 100
  IFNγ and CXCL-9 in serum samples
HSCT cohort: Relationship between IFNγ and the occurrence of GVHD | Day (-7) to day 100
  IFNγ and CXCL-9 in serum samples
IHSCP cohort: IFNγ signature pre-transplant | Day 1
  IFNγ, CXCL-9 and exploratory biomarkers in serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Regis Peffault de Latour, MD, Principal Investigator — Hôpital Saint Louis Paris
Locations (25):
- Belgium (2):
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Roeselare, West-Vlaanderen
  - Cliniques Universitaires Saint-Luc, Brussels
- France (12):
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche, Auvergne-Rhône-Alpes
  - Hôpital Côte De Nacre, Caen, Basse-Normandie
  - Hôpital Pontchaillou, Rennes, Brittany Region
  - Centre Hospitalier Régional et Universitaire de Besançon - Hôpital Jean-Minjoz, Besançon, Franche-Comte
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Centre Hosptitalier Universitaire d'Angers, Angers, Maine Et Loire
  - Hôpital Haut-Lévêque, Pessac, Nouvelle-Aquitaine
  - Hôpital Saint-Eloi, Montpellier Cedex 5, Provence-Alpes-Côte d'Azur Region
  - Hôpital Arnaud de Villeneuve, Montpellier, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Rhône
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hôpital Universitaire Robert-Debré, Paris, Île-de-France Region
- Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg, Germany
- Italy (6):
  - Ospedale Pediatrico Bambino Gesù - Roma - Gianicolo, Roma, Lombardy
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Instituto Giannina Gaslini, Genova
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Regina Margherita, Torino
- Prinses Maxima Centrum Kinderoncologie, Utrecht, Netherlands
- United Kingdom (3):
  - Cardiff and Vale University Health Board, Cardiff, Wales
  - The Royal Marsden Hospital - London, London
  - Imperial College Healthcare NHS Trust NHS Trust, London